CLINICAL TRIAL: NCT04049786
Title: Impact of Roux-en-Y Gastric Bypass (RYGB) Bariatric Surgery on System Pharmacology: Single-dose Cross-over Pharmacokinetic Study of Simvastatin and Carvedilol.
Brief Title: Impact of Bariatric Surgery on Pharmacokinetic Study of Simvastatin and Carvedilol
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Natalia Valadares de Moraes (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); University of Sao Paulo (Other)
Responsible Party: Sponsor-Investigator, Natalia Valadares de Moraes, Assistant Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Organization: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RYGB_pk
Record Dates: First submitted 2019-06-29; First posted 2019-08-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Obesity; Bariatric Surgery; Roux-en Y Gastric Bypass
Keywords: Bariatric surgery; Pharmacokinetics; RYGB; CYP2D6; CYP3A4
MeSH Terms: conditions — Obesity | interventions — Carvedilol; Metoprolol; Simvastatin; Midazolam; Genotype

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Simvastatin - Healthy volunteers (Active Comparator): Adult patients (18-65 years old) with body mass index < 25 kg/mˆ2 treated with a single oral dose of 40 mg simvastatin for Pk analysis. Blood samples collected for blood tests, genomics and transcriptomic analysis
  Interventions: Procedure: Serial blood sampling for PK analysis; Drug: Metoprolol 100 mg for CYP2D6 phenotyping; Drug: Simvastatin 40mg; Drug: Midazolam 2 mg for CYP3A4 phenotyping; Other: Genotyping
- Carvedilol Study - Healthy volunteers (Active Comparator): Adult patients (18-65 years old) with body mass index < 25 kg/mˆ2 treated with a single oral dose of 25 mg carvedilol for Pk analysis. Blood samples collected for blood tests, genomics and transcriptomic analysis
  Interventions: Drug: Carvedilol 25mg; Procedure: Serial blood sampling for PK analysis; Drug: Metoprolol 100 mg for CYP2D6 phenotyping; Drug: Midazolam 2 mg for CYP3A4 phenotyping; Other: Genotyping
- Simvastatin - Obese (Active Comparator): Adult patients (18-65 years old) with body mass index > 30 kg/mˆ2 treated with a single oral dose of 40 mg simvastatin for Pk analysis. Blood samples collected for blood tests, genomics and transcriptomic analysis.
  Interventions: Procedure: Digestive biopsy; Procedure: Serial blood sampling for PK analysis; Drug: Metoprolol 100 mg for CYP2D6 phenotyping; Drug: Simvastatin 40mg; Drug: Midazolam 2 mg for CYP3A4 phenotyping; Other: Genotyping
- Carvedilol study - Obese (Active Comparator): Adult patients (18-65 years old) with body mass index > 30 kg/mˆ2 treated with a single oral dose of 25 mg carvedilol for Pk analysis. Blood samples collected for blood tests, genomics and transcriptomic analysis.
  Interventions: Procedure: Digestive biopsy; Drug: Carvedilol 25mg; Procedure: Serial blood sampling for PK analysis; Drug: Metoprolol 100 mg for CYP2D6 phenotyping; Drug: Midazolam 2 mg for CYP3A4 phenotyping; Other: Genotyping
- Simvastatin - Post-RYGB (Active Comparator): Adult patients (18-65 years old) previously submitted to RYGB surgery treated with a single oral dose of 40 mg simvastatin for Pk analysis. Blood samples collected for blood tests, genomics and transcriptomic analysis.
  Interventions: Procedure: Digestive biopsy; Procedure: Serial blood sampling for PK analysis; Drug: Metoprolol 100 mg for CYP2D6 phenotyping; Drug: Simvastatin 40mg; Drug: Midazolam 2 mg for CYP3A4 phenotyping; Other: Genotyping
- Carvedilol - Post-RYGB (Active Comparator): Adult patients (18-65 years old) previously submitted to RYGB surgery treated with a single oral dose of 25 mg carvedilol for Pk analysis. Blood samples collected for blood tests, genomics and transcriptomic analysis.
  Interventions: Procedure: Digestive biopsy; Drug: Carvedilol 25mg; Procedure: Serial blood sampling for PK analysis; Drug: Metoprolol 100 mg for CYP2D6 phenotyping; Drug: Midazolam 2 mg for CYP3A4 phenotyping; Other: Genotyping

INTERVENTIONS:
Procedure: Digestive biopsy — All patients with indication for RYGB bariatric surgery undergo to endoscopy before and after the surgery as standard protocol. Digestive biopsy are being performed in obese and post-RYGB patients for transcriptomic analysis
  Arms: Carvedilol - Post-RYGB; Carvedilol study - Obese; Simvastatin - Obese; Simvastatin - Post-RYGB
Drug: Carvedilol 25mg — Single-dose of carvedilol 25 mg are being administrated orally.
  Arms: Carvedilol - Post-RYGB; Carvedilol Study - Healthy volunteers; Carvedilol study - Obese
Procedure: Serial blood sampling for PK analysis — Serial blood samples are being collected at times 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15, 18 and 24 hours after drug administration for PK evaluation .
Drug: Metoprolol 100 mg for CYP2D6 phenotyping — Metoprolol is being used as probe drug to evaluate CYP2D6 activity. Single-dose of metoprolol 100 mg are being administrated orally.
Drug: Simvastatin 40mg — Single-dose of simvastatin 40 mg are being administrated orally.
  Other Names: SVA
  Arms: Simvastatin - Healthy volunteers; Simvastatin - Obese; Simvastatin - Post-RYGB
Drug: Midazolam 2 mg for CYP3A4 phenotyping — Midazolam is being used as probe drug to evaluate CYP3A4 activity. Single-dose of midazolam 2 mg are being administrated intravenous.
  Other Names: MDZ
Other: Genotyping — Patients are being genotyped for the main SNP on CYP2C9, ABCB1, SLCO1B1 and CYP2D6 genes using blood samples

SUMMARY:
Obesity affects more than 1 in 3 adults in the U.S. It is commonly associated with reduced quality of life and complications such as metabolic syndrome, heart disease, high blood pressure and sleep disorders. The gastric bypass, also known as Roux-en-Y gastric bypass (RYGB), is one of the most common weight-loss surgeries due to the reliable and long-lasting weight loss and the effective remission of obesity-associated conditions. Although the impact of obesity on absorption, distribution, metabolism and excretion has been documented for several drugs, label recommendations might not account for specific population subgroups, specially morbidly obese patients and obese patients post-bariatric surgery. This study aims to investigate the impact of obesity and RYGB surgery on the kinetic disposition of simvastatin (Study A) and carvedilol (Study B).

DETAILED DESCRIPTION:
The study is ongoing and eligible subjects are enrolled after signing a written informed consent. Research participants (n=120, in total) include healthy volunteers [body mass index (BMI) ≤ 25 kg/m2], obese [BMI > 30 kg/m2] and patients that underwent RYGB surgery 6-60 month prior this research protocol. On day 1, participants receive a single oral dose of 40 mg simvastatin (Study A) or 25 mg racemic carvedilol (Study B). Serial blood samples are collected up to 24 h for the pharmacokinetic analysis. Blood tests (blood count, fasting blood glucose, lipid profile, serum creatinine, urea, gamma-glutamyl transferase, aspartate aminotransferase and alanine amino transferase) are being monitored for all enrolled participants. Blood samples are also collected for genotyping the main genetic polymorphisms associated with carvedilol or simvastatin pharmacokinetics. Metoprolol is being used as a probe drug for CYP2D6 in vivo phenotyping only for research participants enrolled in Study B. After oral administration of metoprolol (on day 2), urine samples are being collected up to 8h after drug administration to determine the urinary metabolic ratio α-hydroxy metoprolol/metoprolol. As part of the pre-surgery evaluation (obese group) or post-surgery follow-up (RYGB group), obese patients and patients post-RYGB are submitted to digestive endoscopies. Healthy participants will not undergo endoscopic examination. The preparation protocol for digestive endoscopy includes: a) 8-hour fasting; b) 10% spray lidocaine (topical); c) oral simethicone (75 mg/ml, 80 drops); d) oxygen therapy depending on the patient (nasal catheter with O2 at 3 L/min); e) 0.02 to 0.03 mg/kg intravenous midazolam; f) 50 mg pethidine. A blood sample is collected 4-h after intravenous midazolam for in vivo CYP3A4 phenotyping. During the endoscopies, duodenum and jejunum biopsies are being collected to investigated interindividual variability related to drug oral bioavailability (only obese and post-RYGB research participants). Samples collected from digestive biopsies will be used to develop individual enteroid microfluidic systems. In vivo phenotyping of drug metabolizing enzymes and transporters will also be assessed by transcriptome using blood samples. The generated in vitro and in vivo data will be combined to build up physiologically based pharmacokinetic models for precision dosing in obese and post-RYGB patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both gender with 18 to 65 years old.
* Healthy volunteers group: body mass index lower or equal to 35 kg/mˆ2.
* Obese group: body mass index higher than 30 kg/mˆ2.
* Post-RYGB group: patients previously submitted to Roux-en-Y gastric bypass bariatric surgery (6-48 months before the study).

Exclusion Criteria:

* Pregnant and lactating patients.
* Patients with serum creatinine higher than 1,5 mg/dL.
* Patients with previous altered coagulation.
* Patients with previous cancer history (on the last year).
* Patients with previous hypersensitivity history to simvastatin or carvedilol.
* Patients who were in use of any anticoagulant (heparin, low molecular weight heparin, aspirin, nonsteroidal antiinflammatory drugs).
* Patients who were in use of CYP3A4 or P-glycoprotein inhibitors or inducers.
* For carvedilol study: patients who were in use of CYP2D6 inhibitors; poor metabolizer phenotype of CYP2D6 and genotyped as CYP2C9*3/*3.
* Patients who disagree to continue the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic analysis of simvastatin | Time 0 up to 24 hours after single dose simvastatin administration.
  Population pharmacokinetic modeling and simulation.
Pharmacokinetic analysis of carvedilol | From time 0 up to 24 hours after single dose carvedilol administration
  Population pharmacokinetic modeling and simulation.

SECONDARY OUTCOMES:
CYP2D6 phenotyping using metoprolol as a probe drug | Urine sampling collected from time 0 up to 8 hours after metoprolol administration
  The CYP2D6 phenotype was determined by urinary concentration ratio metoprolol/alfa-hydroxymetoprolol.
CYP3A4 phenotyping using midazolam as a probe drug | Day 2: a blood sample will be collected after midazolam administration
  Midazolam plasma concentration will be determined by chromatographic analysis
Genotyping the main SNPs on CYP2C9, CYP2D6, ABCB1 and SLCO1B1 genes | Day 1: a blood sample will be collected immediately after your check-in in the clinical research unit
  The main SNPs on CYP2C9, CYP2D6, ABCB1 and SLCO1B1 genes will be evaluated by RT-PCR
Transcriptomic analysis of liver extracellular vesicles | Day 1: a blood sample will be collected immediately after your check-in in the clinical research unit
  Expression levels of transporters and enzymes will be quantified by real-time quantitative PCR
Transcriptomic analysis of intestine samples | Digestive biopsy collected in the second day of research protocol
  Expression levels of transporters and enzymes will be quantified by real-time quantitative PCR

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Salgado Junior, PhD, Principal Investigator — University of Sao Paulo; Jose S dos Santos, PhD, Principal Investigator — University of Sao Paulo; Natalia De Moraes, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Orlando, Florida, United States